CLINICAL TRIAL: NCT03217344
Title: Conservative Treatment of Proximal Humeral Fractures - Immobilization for 1 Week Compared to Three Weeks: Prospective Randomized Study
Brief Title: Conservative Treatment of Proximal Humeral Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Carlos Torrens, Medical Doctor, Hospital del Mar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016/6588/I
Record Dates: First submitted 2017-07-04; First posted 2017-07-14 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Shoulder Fractures
MeSH Terms: conditions — Shoulder Fractures | interventions — Conservative Treatment

STUDY DESIGN:
Intervention Model Description: prospective randomized without restrictions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1-week (Experimental): patients undergoing 1-week immobilization period
  Interventions: Procedure: conservative treatment
- 3-week (Experimental): patients undergoing 3-week immobilization period
  Interventions: Procedure: conservative treatment

INTERVENTIONS:
Procedure: conservative treatment — immobilization on sling of the injured arm

SUMMARY:
Optimal treatment of proximal humeral fractures is yet to be defined. Many of them can be treated non-operatively. The question remains on how long do we have to immobilize non-operatively treated proximal humeral fractures?

DETAILED DESCRIPTION:
There is still controversy on best treatment of proximal humeral fractures. While some authors propose surgical treatment other advocate for conservative treatment. Traditionally, fractures treated non-operatively undergo a 3-week period of immobilization followed by progressive rehabilitation program. Nevertheless, there is little evidence to support a 3-week immobilization period. The purpose of this study is to bring evidence to support either a 1-week immobilization or 3-week immobilization period in non-operatively treated proximal humeral fractures.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 60 yo and < 85 yo
* Acute fractures less than 1 week evolution
* Conservative treatment decided by orthopedic surgeon
* Contact between humeral head and humeral shaft.
* No gleno-humeral dislocation
* No previous surgery

Exclusion Criteria:

* Cognitive impairment

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
pain (analogical pain scale) | 1 year
  pain assessment through all the follow-up through the analogical pain scale

SECONDARY OUTCOMES:
fragment displacement assessed through X-Ray exam | 3 months
  displacement of the fractured fragments within 3 months period assessed through X-Ray exam
functional outcome | 1 year
  functional outcome measured through Constant Score

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Torrens, PhD, Principal Investigator — Hospital Mar
Locations (1):
- Carlos Torrens, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196